CLINICAL TRIAL: NCT05353959
Title: Progression of Prodromal Markers of α-synucleinopathy Neurodegeneration in the First-degree Relatives of Patients With REM Sleep Behavior Disorder: a 7-year Prospective Study
Brief Title: Progression Follow up of the First-degree Relatives of Patients With REM Sleep Behavior Disorder
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Wing Yun Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: RGC14116121
Record Dates: First submitted 2021-12-21; First posted 2022-04-29 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Neurodegeneration; Prodromal markers; REM sleep behavior disorder
MeSH Terms: conditions — Parkinson Disease; Nerve Degeneration; REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
REM sleep behavior disorder is a novel and distinct parasomnia characterized by recurrent dream enactment behaviors (DEBs) and polysomnographic features of REM sleep without atonia (RSWA), with typical onset age at early 60's. Idiopathic RBD (iRBD) has been suggested as a most specific precursor of α-synucleinopathy-related neurodegeneration (e.g. Parkinson's disease (PD)). There are increasing reports of positive familial cases in both iRBD and PD. In the past few years, the investigators have established the baseline data of a case-control family cohort of iRBD (208 first-degree relatives (FDR) of patients with iRBD and 204 FDRs of controls). Not only did the investigators confirm the familial aggregation of iRBD with neurodegeneration and iRBD cases, the investigator also found that the FDRs harbored a spectrum of isolated RBD features (including DEBs, REM- sleep behavioral events, and RSWA). Besides, when compared with control-FDRs, iRBD-FDRs patients showed more prodromal markers of neurodegeneration (including possible/probable RBD, excessive daytime sleepiness, constipation, and subthreshold parkinsonism) as suggested by the International Parkinson and Movement Disorder Society (MDS) research criteria. The promising baseline findings paved the way for the current proposed prospective study of this unique family cohort. In addition, around 85 unaffected FDRs from each group has repeated the assessments at a mean follow-up duration of about 4 years (early termination of the study supported by RGC- ECS Ref no. 24117018; reason for early termination - ECS PI applicant left the University at early 2020), the preliminary data indicated a persistent familial aggregation of RBD symptoms, loading of prodromal markers (e.g. possible RBD, subthreshold parkinsonism), and a seemingly faster progression into prodromal RBD among the FDRs of iRBD than that of control. This current proposed study is a prospective study with a mean of 7-year follow-up interval to monitor the progression of α- synucleinopathy neurodegeneration and related markers. With the rolling recruitment, the investigators now have 230 control-FDRs and 250 iRBD-FDRs, from which the investigators expect 200 FDRs of each group may respond to the follow-up study. A series of prodromal markers related to neurodegeneration including clinical and sleep assessment (e.g. autonomic symptoms, motor signs, neurocognitive function, sleepiness, vPSG and one-week actigraphy) that were measured at baseline will be reassessed. Specifically, home PSG with a body-movement monitoring system will be additionally implemented in the proposed study to empower the identification of RBD features, especially during the COVID pandemic period at which hospital accessibility is restricted. In addition, the development of clinical neurodegenerative diseases will be ascertained. This proposed study, by recruiting FDRs of iRBD patients (and controls) with prospective study design, will provide novel and important information on the progression of prodromal makers of α-synucleinopathy neurodegenerative diseases in a high-risk population and facilitate further genetic/omics and future neuroprotective intervention study of the familial iRBD.

DETAILED DESCRIPTION:
Idiopathic RBD (iRBD) as a specific prodromal marker of α-synucleinopathy Rapid eye movement (REM) sleep behavior disorder (RBD) is a parasomnia characterized by abnormal behavioral manifestations and the loss of muscle atonia during REM sleep (i.e. REM sleep without atonia, RSWA). Accumulating evidence suggests that iRBD is an integral part of the progression of α-synucleinopathy neurodegeneration, including Parkinson's disease (PD), dementia with Lewy bodies, and multiple system atrophy. A recent meta-analysis has summarized that over 95% of patients with iRBD would eventually develop neurodegenerative diseases after 14 years of follow-up. Patients with iRBD have an increased prevalence of other non-motor symptoms (or prodromal markers) closely related to PD, including autonomic dysfunction, olfactory loss, color vision impairment, neurocognitive impairment, neuroimaging of dopamine dysfunction, daytime sleepiness, and psychiatric disorders. Furthermore, a series of studies have found that these markers might confer a higher risk of developing future neurodegenerative diseases in patients with iRBD. The integration of these risk factors and biomarkers could greatly improve the predictive value of future neurodegeneration. In this regard, the International Parkinson and Movement Disorder Society (MDS) proposed research criteria for prodromal PD in 2015 (and had an update in 2019). The MDS research criteria combine estimates of background risk (environmental risk factors and genetic findings) and results of diagnostic marker testing to estimate the probability of prodromal PD.

According to the MDS criteria, PSG-confirmed iRBD possesses the highest likelihood ratio of the probability of PD (positive likelihood ratio of 130) among all risk factors and biomarkers. In other words, iRBD is the ideal model in which all these risk factors and biomarkers related to neurodegeneration can be tested in prospective studies. Indeed, a recent study has found that 74% of iRBD patients met the MDS criteria for probable prodromal Parkinson's compared to 0.3% of controls. One recent prospective study has further supported that the MDS research criteria for prodromal PD as a promising indicator to predict the new incidence of α-synucleinopathy in patients with iRBD. The concept of prodromal RBD refers to the cases when patients presented with isolated RSWA (without typical nocturnal behavioral manifestations), or isolated REM-sleep-related behavioral events (including typical dream-enactment behaviors that are assumed to occur in REM sleep), and a definite diagnosis of RBD could not be confirmed, but instead, a prodromal phase of RBD is suggested.10 Limited studies including our data (manuscript in submission) have suggested that even patients with prodromal RBD are associated with a higher risk for neurodegeneration than controls. Thus, identification of prodromal RBD helps early detection of the individuals at risk for neurodegeneration for future disease-modifying trials. However, it is not clear on whether any specific prodromal markers will progress in the prodromal stage of RBD, and whether the occurrence of the prodromal stage is associated with any risk factors. Thus, it is necessary to prospectively investigate the prodromal RBD and associated markers in a group of people at risk for RBD, for example, the unaffected relatives of the familial RBD.

A few studies have tried to document the progression and evolution of risk factors and prodromal markers of PD in healthy subjects, at-risk individuals, and patients with early PD. It has been shown that the percentage of mentalis tonic EMG activity, a predictor of the development of neurodegenerative diseases in iRBD, significantly increases from 30% to 54% in patients with iRBD after 5 years. A recent 2-year prospective study examining the progression of 30 markers related to early PD has found that sleep problems, non-motor symptoms, and imaging measures significantly change with time and may serve as informative markers to quantify the progression of PD. It has also been shown that individuals at risk of PD (e.g. GBA mutation carriers) may present with a faster progression of some prodromal markers of early PD over time than healthy controls. In these regards, monitoring the progression of prodromal markers among at-risk individuals (such as individuals with a positive family history of RBD) is pertinent, which may help to map the disease course from prodromal to syndromal phase.

There are some knowledge gaps regarding familial aggregation and progression of prodromal markers of PD in iRBD. First, although the investigators have confirmed the familial aggregation of iRBD, the mean age of FDRs (around 54 years) at baseline was relatively younger than the typical age onset of iRBD (around 60 years). The timely follow-up at around 7-year interval will be at the perfect timing to detect the familial aggregation of RBD and its core features as the clinical phenotype related to iRBD may not have emerged in the younger-aged population (e.g. offspring) at baseline. It is reasonable to expect a higher rate of definite iRBD as confirmed by vPSG (including home PSG monitoring system) in the FDRs and a stronger familial aggregation in this 7-year prospective follow-up. Second, although a few prospective studies have suggested the progression of some prodromal makers of early PD in iRBD, there is a lack of study in FDRs of iRBD patients. It is unclear whether iRBD-FDRs also present with a more rapid progression of these potential neurodegenerative markers in terms of frequency and severity, which might predict the onset of definite RBD and neurodegenerative diseases. In these regards, prospective studies with a regular and adequate duration of follow-up are needed to optimally map the progression and evolution of prodromal markers, onset of RBD, and neurodegenerative diseases. Finally, other markers (such as physical activity and circadian rhythm and tonic EMG activity level), albeit not being included in the MDS research criteria for Prodromal PD, are reliably associated with PD or other neurodegenerative diseases. In this regard, it is also interesting to investigate whether these indicators will additionally predict the progression of PD and related markers.

ELIGIBILITY:
Inclusion Criteria:

* Chinese aged 40 or above
* Can give informed consent for participation in the study
* Sex- and age matched between groups

Exclusion Criteria:

* younger than 40
* not capable of giving informed consent for participation in the study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The total number of FDRs for face-to-face interview would be 200 for each group
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-01-02 (Estimated)

PRIMARY OUTCOMES:
Parkinson's disease | 7 years
  Number of participants with progression to Parkinson's disease based on the MDS research criteria for prodromal Parkinson's disease

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kwok Wing, Prof, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Shatin Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided